CLINICAL TRIAL: NCT00459849
Title: Tilting of Radioactive Plaques After Initial Accurate Placement for Treatment of Uveal Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barnes Retina Institute (Other)
Responsible Party: Archavan Almony, M.D., Barnes Retina Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRPO# 07-0092
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Uveal Melanoma
Keywords: Melanoma; Brachytherapy; Ultrasonography
MeSH Terms: conditions — Uveal Melanoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intraoperative ultrasonography — Intraoperative ultrasonography will be used to determine plaque placement.

SUMMARY:
Plaque radiotherapy is a common treatment for uveal melanoma. However, local failure has been reported in up to 20% of patients. We use intraoperative ultrasonography at plaque insertion and removal to evaluate plaque movement as a potential factor in local failure.

DETAILED DESCRIPTION:
Episcleral plaque radiotherapy is a common treatment for uveal melanoma and results in local tumor control in most cases. However, local failure has been reported in a substantial proportion of patients. Since local failure greatly increases the risk of metastatic death, identifying and correcting the causes of local treatment failure are of paramount importance. Poor plaque localization is an important contributing factor to local failure. With the aid of intraoperative ultrasonography, most malpositioned plaques can be identified and readjusted at the time of plaque insertion. However, little is known about plaque movement during the 4-5 days of brachytherapy, which could also contribute to local failure. To address this question, we perform intraoperative B-scan ultrasonography at the time of iodine-125 radioactive plaque insertion and removal in uveal melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with uveal melanoma treated with brachytherapy

Exclusion Criteria:

* Ciliary melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2000-07; Primary Completion 2007-07 (Estimated); Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Plaque tilt using intraoperative ultrasonography | End of study
Local melanoma failure | End of study

CONTACTS AND LOCATIONS:
Overall Officials: J W Harbour, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Harbour JW. Clinical overview of uveal melanoma: introduction to tumors of the eye. In: Albert DM, Polans A, eds. Ocular Oncology. New York: Marcel Dekker; 2003:1-18.
- [Background] Char DH, Quivey JM, Castro JR, Kroll S, Phillips T. Helium ions versus iodine 125 brachytherapy in the management of uveal melanoma. A prospective, randomized, dynamically balanced trial. Ophthalmology. 1993 Oct;100(10):1547-54. doi: 10.1016/s0161-6420(93)31446-6. PMID 8414414
- [Background] Garretson BR, Robertson DM, Earle JD. Choroidal melanoma treatment with iodine 125 brachytherapy. Arch Ophthalmol. 1987 Oct;105(10):1394-7. doi: 10.1001/archopht.1987.01060100096035. PMID 3310986
- [Background] Karlsson UL, Augsburger JJ, Shields JA, Markoe AM, Brady LW, Woodleigh R. Recurrence of posterior uveal melanoma after 60Co episcleral plaque therapy. Ophthalmology. 1989 Mar;96(3):382-8. doi: 10.1016/s0161-6420(89)32882-x. PMID 2710530
- [Background] Quivey JM, Augsburger J, Snelling L, Brady LW. 125I plaque therapy for uveal melanoma. Analysis of the impact of time and dose factors on local control. Cancer. 1996 Jun 1;77(11):2356-62. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-V. PMID 8635107
- [Derived] Almony A, Breit S, Zhao H, Garcia-Ramirez J, Mansur DB, Harbour JW. Tilting of radioactive plaques after initial accurate placement for treatment of uveal melanoma. Arch Ophthalmol. 2008 Jan;126(1):65-70. doi: 10.1001/archophthalmol.2007.9. PMID 18195220